CLINICAL TRIAL: NCT00973518
Title: Improved Diagnosis of Alzheimer's Disease Using Magnetoencephalography (MEG) and the Synchronous Neural Interaction Test: A One-month Study
Brief Title: Improved Diagnosis of Alzheimer's Disease Using Magnetoencephalography (MEG)
Status: Completed | Type: Observational
Sponsor: Orasi Medical, Inc. (Industry)
Responsible Party: Todd Verdoorn, Ph.D., Chief Scientific Officer, Orasi Medical, Inc.
Other Study IDs: ADD 09-02
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; AD; Healthy Control
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alzheimer's Disease subjects: Subjects diagnosed with dementia of Alzheimer's type (DSM-IV-TR).
- Healthy Control subjects: Age & gender-matched subjects determined to be healthy.

SUMMARY:
The current study is intended to enrich and extend the database of Alzheimer's Disease (AD) and healthy control (HC) MEG scans and will include patients meeting DSM-IV-TR criteria for dementia of Alzheimer's type, and age- and gender-matched HC subjects meeting criteria of normal neurological function. This study will include 2 MEG and electroencephalography (EEG) scans on approximately 80 AD subjects and 80 HC subjects over approximately 30 days. All subjects will have MEG/EEG scans at baseline and 28 - 35 days after baseline. Within one day of each scan visit AD subjects will undergo 4 standard functional tests while HC subjects will undergo 2 standard functional tests.

This study will test the following hypotheses:

* MEG scans of resting-state, eyes-open brain function reveal patterns of correlated activity that differ between HC subjects and subjects diagnosed with dementia of Alzheimer's type;
* Patterns of correlated activity measured in AD subjects correspond to other measures of disease severity such as standard functional test scores;
* MEG scan patterns for HC subjects are consistent across repeated measures taken over a 30 day period.

DETAILED DESCRIPTION:
This study is intended to extend the capabilities of the Synchronous Neural Interaction® (SNI) test, which is under development by the sponsor, Orasi Medical, Inc. Magnetoencephalography (MEG) is an FDA-approved, non-invasive technique used to measure magnetic fields generated by small intracellular electrical currents in neurons. The SNI test evaluates brain function and dysfunction by analyzing brief (1 minute) MEG scans and comparing individual scan results to a database of MEG scans and clinical information. Proprietary software algorithms process the data generated by MEG instruments allowing Orasi to use the SNI test for accurate tracking and diagnosis of neurological disorders such as Alzheimer's disease (AD) and Multiple Sclerosis (MS). The current study is intended to enrich and extend the database of AD and healthy control (HC) MEG scans and will include patients meeting DSM-IV-TR criteria for dementia of Alzheimer's type, and age- and gender-matched HC subjects meeting criteria of normal neurological function. This study will include 2 MEG and EEG scans on approximately 80 AD subjects and 80 HC subjects over approximately 30 days. All subjects will have MEG/EEG scans at baseline and 28 - 35 days after baseline. Within one day of each scan visit AD subjects will undergo 4 standard functional tests while HC subjects will undergo 2 standard functional tests. The results generated in this study will be used to improve the accuracy of the SNI test for diagnosing and tracking the progression of AD. Once a robust training set or template is described, Orasi Medical will conduct additional clinical studies to formally test the diagnostic accuracy of the technology and support applications for regulatory approval to market the SNI test for AD. The objective of this work is to produce and validate a novel tracking and diagnostic technology for AD that is more selective and sensitive than currently available diagnostic tools.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with dementia of Alzheimer's type (DSM-IV-TR) or is serving as a healthy control subject with normal neurological function based on medical history and following neurological exam.
* AD Subject has a screen MMSE raw score > 16 or HC subject has a screen MMSE raw score > 26.
* Subject is between 50 and 90 years of age at the time of screening.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is a non-smoker.
* Subject is judged to be in good health other than AD, based on medical history and brief physical examination.
* AD subject has a care-giver or spouse who is willing and able to assure subject compliance with study procedures or subject is participating as a healthy control subject.

Exclusion Criteria:

* Subject has a history or diagnosis of a significant neurological condition other than Alzheimer's disease including Parkinson's disease, vascular dementia, Lewy body dementia, frontal temporal dementia, human immunodeficiency virus, multiple sclerosis, seizures, epilepsy, stroke, ADHD, dyslexia, or severe traumatic brain injury.
* Subject has a history of primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, delusional disorder) or bipolar disorder.
* Subject has a Modified Hachinski Ischemia Scale (HIS) score greater than 4.
* The subject has a recent history (within 2 years) of alcohol or substance abuse/dependence.
* Subject had an MRI within two weeks prior to Study Day 1.
* Subject has metal dental braces, pacemaker or other common medical devices that may interfere with the MEG scan.
* Subject is unable to complete the MEG scan procedure.
* Investigator has any concern regarding the safe participation of a subject in the study, or if for any other reason the investigator considers the subject inappropriate for study participation.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The current study will include patients meeting DSM-IV-TR criteria for dementia of Alzheimer's type, and age- and gender-matched healthy control subjects meeting criteria of normal neurological function.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of patterns of correlated brain activity measured by MEG and the Orasi SNI test that differ consistently (e.g. at all evaluation time points) between HC and AD subjects | approximately 30 days
Identification and characterization of patterns of correlated brain activity measured by MEG and the Orasi SNI test that differ across time points within single subjects and across groups of HC and AD subjects | Approximately 30 days

SECONDARY OUTCOMES:
Identification and characterization of Orasi SNI test features that correlate with independent measures of cognitive function based on functional testing (ADAS-Cog sum of boxes, and MMSE raw score, One Card Learning Test) | Approximately 30 days
Identification and characterization of Orasi SNI test features that correlate with AD medications being taken by AD subjects | Approximately one month
Identification, characterization and comparison of scan results generated by MEG and EEG | Approximately one month

CONTACTS AND LOCATIONS:
Overall Officials: Concetta Forchetti, MD, PhD, Principal Investigator — Alexian Brothers Neuroscience Institute; Raj C Shah, MD, Principal Investigator — Rush Alzheimer's Disease Center
Locations (2):
- United States (2):
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois